CLINICAL TRIAL: NCT04798456
Title: A Multimodal Approach to Personalized Tracking of Evolving State-Of-Consciousness in Brain- Injured Patients
Brief Title: Aiming for a Better Understanding and Improvement of the Diagnosis and Prognosis of Patients With Disorders of Consciousness Through Multimodal Observations
Acronym: PerBrain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Brain Institute (ICM) (Other)
Collaborators: University of Milan (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Weizmann Institute of Science (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Jacobo Sitt, Research Director, INSERM, Paris Brain Institute (ICM)
Other Study IDs: ERAPERMED2019-101 - PerBrain; 01KU2003 (Other Grant/Funding Number: Federal ministry for education and research (Germany))
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Disorders of Consciousness; Minimally Conscious State; Unresponsive Wakefulness Syndrome; Caregivers
Keywords: Clinical Neuroscience; Disorders of Consciousness; Neuroimaging; Brain-Body interactions; Multimodal precision diagnosis; Machine Learning; Caregivers well-being; Unresponsive wakefulness syndrome; Minimally conscious state
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Diagnostic Imaging; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with DoC
  Interventions: Behavioral: Coma scales; Diagnostic Test: Imaging, electrophysiology, body signals, and brain stimulation
- Caregivers/ legal guardian of patients with DoC
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Coma scales — CRS-R and GOSE
  Groups: Patients with DoC
Diagnostic Test: Imaging, electrophysiology, body signals, and brain stimulation — MRI, fMRI, EEG, TMS-EEG, Olfaction, Respiration, EKG
  Groups: Patients with DoC
Behavioral: Questionnaires — several questionnaires and an interview with the caregiver
  Groups: Caregivers/ legal guardian of patients with DoC

SUMMARY:
Improved treatment of severe brain injuries has resulted in increased survival rates. While some of these patients regain consciousness after a transient state of coma, others may develop a disorder of consciousness (DoC). Diagnosis of DoC currently relies on standardized behavioral assessment. The importance of accuracy in such diagnosis cannot be overstated, as it guides critical decisions on treatment (including pain management), and could underlie end-of-life decisions. Despite this importance, current behavioral diagnosis often fails, if because of the major sensory and motor deficits associated with DoC, or because of the heterogeneous etiology and pathophysiology associated with the condition. Finally, the need for accurate diagnosis and prognosis transcends the needs of the patients alone: caregiving of these patients is very stressful, principally for the large uncertainty associated with them. Thus, more accurate diagnosis and prognosis provide major relief for caregivers, and paradoxically, even if the news is not "good". For all these reasons it is critical to developing personalized diagnosis and prognosis prediction tools that permit a stratified analysis at the single-patient level. The PerBrain Project will benefit from the multidisciplinary partners' expertise, and the unique opportunity to perform longitudinal assessments in four clinical sites through both established and novel electrophysiological, neuroimaging, and physiological techniques. Based on the collected data, the investigators will develop a multimodal personalized diagnostic tool for DoC patients using state-of-the-art computational tools, such as machine learning, in order to better determine the current state (diagnosis) and future outcome (prognosis). The overall aim of this project will provide for a better understanding of the pathophysiological mechanisms in DoC, which will, in turn, allow personalized rehabilitation strategies, and improved single-patient predictions of state and prognosis.

ELIGIBILITY:
* Recruitment is taking place in:

  * France, Paris, Pitie-Salpetriere Hospital;
  * Italy, Milan, Dipartimento di Cura e Riabilitazione delle Gravi Cerebrolesioni Acquisite (GCA);
  * Israel, Raanana, Loewenstein Hospital;
  * Germany, Munich: intensive care units of the University Clinic LMU Munich and Therapiezentrum Burgau
* Inclusion criteria:

  * Disorder of consciousness (UWS and MCS) patients and their caregiver/legal guardian
  * Patient age: 18-85 years
  * Informed consent signed by legal guardian
* Exclusion criteria:

  * Pregnancy
  * Pre-existing coma/VS/MCS
  * Continuous medical sedation (induced coma)
  * Use of barbiturates for sedation
  * Terminal malignant disease, as it increases the likelihood of not being alive for the 12-month follow-up
  * Prediction of a highly unlikely survival until the time of the 12-month follow-up due to conditions such as multi-organ failure based on the judgement of a critical care physician
  * Withdrawal of life-support
  * Palliative care setting
  * Epileptic seizures (TMS contraindication)
  * MRI contraindications (magnetic material in or on person such as pacemakers, cochlear implants, shell splinters, metal plates, certain prosthetic joints/limbs, copper-based intrauterine device, magnetic clips or stents, some large tattoos)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care units and rehabilitation centres
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Patients: Implementation of a hierarchical multi-modal personalized procedure to diagnose and track the change of the state of consciousness in brain-injured patients | Changes from T1: 1-2 Months from injury; T2: 4-7 Months from injury; T3: 9-12 months from injury
  Coma Recovery Scale Revised (CRS-R) [0-23] Higher score better outcome
Patients: Implementation of a hierarchical multi-modal personalized procedure to diagnose and track the change of the state of consciousness in brain-injured patients | Changes from T1: 1-2 Months from injury; T2: 4-7 Months from injury; T3: 9-12 months from injury
  Extended Glasgow Outcome Scale (GOSE) [1-8] Higher score better outcome
Patients: Implementation of a hierarchical multi-modal personalized procedure to diagnose and track the change of the state of consciousness in brain-injured patients | Changes from T1: 1-2 Months from injury; T2: 4-7 Months from injury; T3: 9-12 months from injury
  Quantitative high density EEG (64 Electrodes)
Patients: Implementation of a hierarchical multi-modal personalized procedure to diagnose and track the change of the state of consciousness in brain-injured patients | Changes from T1: 1-2 Months from injury; T2: 4-7 Months from injury; T3: 9-12 months from injury
  Standard EEG and transcranial magnetic stimulation (TMS-EEG)
Patients: Implementation of a hierarchical multi-modal personalized procedure to diagnose and track the change of the state of consciousness in brain-injured patients | Changes from T1: 1-2 Months from injury; T2: 4-7 Months from injury; T3: 9-12 months from injury
  Structural MRI and functional MRI (without contrast agent)
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Sociodemographic characteristics
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Brief Illness Perception Questionnaire (BIPQ) [0-80] Higher score more positive illness representation
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Euro-Qol 5 (EQ-5D61) [0-15] higher values indicating better perceived quality of life.
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from 0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Adult Carer Quality of Life Questionnaire (ACQoL24) [0-120] higher values better quality of life
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Hospital Anxiety and Depression Scale (HADS) [0-52] higher scores indicating higher levels of anxiety and depression.
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Resilience (RS14) [14-98] higher scores relate to higher resilience levels.
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Sense of coherence (SOCS) [13-91] higher scores indicate higher sense of coherence.
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Treatment choices survey [28-140] higher score indicates a stronger agreement with the treatment and higher reason to take a given treatment decision
Caregivers: use of questionnaires to asses change in factors that impact well-being and treatment decisions of informal caregivers/family members confronted with multimodal technology-based tests for DoC patients | Changes from C0: before T1 (1-2 Months from injury); C1: between T1(1-2 Months from injury) and T2 (4-7 Months from injury); C2: between T2 (4-7 Months from injury) and T3 (9-12 Months from injury); C3: after T3 (9-12 Months from injury)
  Semi-structured qualitative Interview based on a thematic grid for brochure development

SECONDARY OUTCOMES:
Caregivers: develop a brochure/guide to be applied in clinical practice for the effective communication of technology-based results | 12 months
  Working closely with Patient organizations/ patient representatives:
  Representatives of organizations ("Schädel- Hirnpatienten in Not e.V." in Germany) will be consulted in focus groups to jointly discuss the met and unmet needs and communication problems reported by caregivers in the study. Additionally, we will conduct a semi-structures interview with the caregivers. This information will help to devise with the research team effective communication strategies to be implemented in a brochure for the presentation of multimodal technology-based DOC testing.

CONTACTS AND LOCATIONS:
Locations (4):
- Paris Brain Institute (ICM), Paris, France
- University Hospital of the Ludwig-Maximilians-University of Munich, Munich, Germany
- Loewenstein Hospital, Raanana, Israel
- Dipartimento di Cura e Riabilitazione delle Gravi Cerebrolesioni Acquisite (GCA), Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacino JT, Kalmar K. Diagnostic and prognostic guidelines for the vegetative and minimally conscious states. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):166-74. doi: 10.1080/09602010443000498. PMID 16350959
- [Background] Raimondo F, Rohaut B, Demertzi A, Valente M, Engemann DA, Salti M, Fernandez Slezak D, Naccache L, Sitt JD. Brain-heart interactions reveal consciousness in noncommunicating patients. Ann Neurol. 2017 Oct;82(4):578-591. doi: 10.1002/ana.25045. Epub 2017 Oct 11. PMID 28892566
- [Background] Arzi A, Rozenkrantz L, Gorodisky L, Rozenkrantz D, Holtzman Y, Ravia A, Bekinschtein TA, Galperin T, Krimchansky BZ, Cohen G, Oksamitni A, Aidinoff E, Sacher Y, Sobel N. Olfactory sniffing signals consciousness in unresponsive patients with brain injuries. Nature. 2020 May;581(7809):428-433. doi: 10.1038/s41586-020-2245-5. Epub 2020 Apr 29. PMID 32461641
- [Background] Casali AG, Gosseries O, Rosanova M, Boly M, Sarasso S, Casali KR, Casarotto S, Bruno MA, Laureys S, Tononi G, Massimini M. A theoretically based index of consciousness independent of sensory processing and behavior. Sci Transl Med. 2013 Aug 14;5(198):198ra105. doi: 10.1126/scitranslmed.3006294. PMID 23946194
- [Background] Engemann DA, Raimondo F, King JR, Rohaut B, Louppe G, Faugeras F, Annen J, Cassol H, Gosseries O, Fernandez-Slezak D, Laureys S, Naccache L, Dehaene S, Sitt JD. Robust EEG-based cross-site and cross-protocol classification of states of consciousness. Brain. 2018 Nov 1;141(11):3179-3192. doi: 10.1093/brain/awy251. PMID 30285102
- [Background] Vogler J, Klein AM, Bender A. Long-term health-related quality-of-life in patients with acquired brain injury and their caregivers. Brain Inj. 2014;28(11):1381-8. doi: 10.3109/02699052.2014.919536. Epub 2014 Jun 19. PMID 24945467
- [Derived] Derchi CC, Comanducci A, Bassi M, Rosenfelder MJ, Valota C, Willacker L, Oehl P, Rosanova M, Sitt JD, Bender A, Kuehlmeyer K. Surrogate decision-making for people with disorders of consciousness: considering the control-preferences of informal caregivers before implementing multimodal testing. BMC Med Ethics. 2026 Jan 2. doi: 10.1186/s12910-025-01357-4. Online ahead of print. PMID 41484601
- [Derived] Willacker L, Raiser TM, Bassi M, Bender A, Comanducci A, Rosanova M, Sobel N, Arzi A, Belloli L, Casarotto S, Colombo M, Derchi CC, Flo Rama E, Grill E, Hohl M, Kuehlmeyer K, Manasova D, Rosenfelder MJ, Valota C, Sitt JD. PerBrain: a multimodal approach to personalized tracking of evolving state-of-consciousness in brain-injured patients: protocol of an international, multicentric, observational study. BMC Neurol. 2022 Dec 9;22(1):468. doi: 10.1186/s12883-022-02958-x. PMID 36494776